CLINICAL TRIAL: NCT02288988
Title: Results of the Minimally Invasive Collis-Nissen Technique for the Treatment of True Short Esophagus
Brief Title: Minimally Invasive Collis-Nissen for the Treatment of Short Esophagus
Acronym: COLLIS-NIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bologna (Other)
Responsible Party: Principal Investigator, Sandro Mattioli, Associate Professor, University of Bologna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Collis-Nissen Surgery
Record Dates: First submitted 2014-11-04; First posted 2014-11-13 (Estimated); Last update posted 2014-11-13 (Estimated); Status verified 2014-11

CONDITIONS: Gastro-esophageal Reflux Diseases; Short Esophagus
Keywords: GERD; Short Esophagus; Minimally Invasive Surgery; Collis gastroplasty
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Gastroplasty; Fundoplication

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- GERD patients with Short Esophagus (Other): Patients with True Short Esophagus diagnosed intra-operatively: The length of the intra-abdominal portion of the esophagus < 2.5 cm measured intra-operatively using a combined endoscopic-laparoscopic method. Minimally invasive antireflux surgery was performed (Collis gastroplasty + Nissen fundoplication).
  Interventions: Procedure: Antireflux Surgery

INTERVENTIONS:
Procedure: Antireflux Surgery — Collis gasytroplasty Nissen antireflux fundoplication
  Other Names: Collis gastroplasty; Nissen

SUMMARY:
True short esophagus (TSE) is present when the distance between the esophago-gastric (E-G) junction and the apex of the hiatus is shorter than 2.5 cm, without the application of any downward pressure on the stomach, after maximal mobilization of the distal thoracic esophagus. It has been demonstrated that TSE is present in 20% of patients undergoing routine surgery for gastro-esophageal reflux disease (GERD), and in more than 50% of cases of type III-IV hiatal hernia (HH) that are treated surgically. Recent reports have confirmed the importance of diagnosing and electively treating TSE to reduce the risk of anatomic recurrence after surgery. The surgical techniques currently used for the elective treatment of TSE are based on the association of the Collis gastroplasty with an anti-reflux funduplication and the hiatoplasty, performed using minimally invasive techniques; the mortality, morbidity, and outcomes of these procedures remain subjects of debate. In light of the doubtful validity of the surgical results for TSE, some researchers have proposed that this condition should not be treated with surgical therapy. In the absence of randomized, multicenter studies designed to compare the surgical techniques used to treat TSE, the investigators believe that data obtained from a single-center study may be useful to the surgical community, provided that such data are based on an objective intra-operative diagnosis of TSE and a rigorous follow-up period.

DETAILED DESCRIPTION:
The pre-operative evaluation included a clinical interview, a barium swallow study, an upper gastro-intestinal (GI) endoscopy, and standard manometry. The type and severity of symptoms and the grade of reflux esophagitis were determined using a questionnaire with semi-quantitative scales.

The barium swallow study was performed to define the position of the E-G junction with respect to the diaphragm with the patient in the upright position, as well as the morphology and the type of HH. The migration of the E-G junction was radiologically diagnosed in three steps using the following differential diagnoses: hiatal insufficiency, concentric HH, and acquired short esophagus. Reflux esophagitis was classified according to the Los Angeles classification. In the absence of grade A esophagitis or a more severe type of esophagitis, patients underwent 24-h pH recording or intraluminal impedance/pH monitoring. The need for surgical therapy was determined according to defined parameters and to the current guidelines for GERD therapy.

The patient is placed in the lithotomic position; the pelvis and left chest are lifted 45° to the right to facilitate access for a left thoracostomy along the posterior axillary line.

Surgery begins via five laparoscopic ports: the camera port is placed 5 to 10 cm above the umbilicus, depending on the patient's body size, to enable access to the upper portion of the mediastinum. After the opening of the phreno-esophageal membrane, the E-G junction is isolated and the sac and fat pad (with the exception of the fat near the lesser curvature to preserve the integrity of the vagus nerves) are resected. A fiber endoscope is inserted trans-orally to determine the position of the upper margins of the gastric folds, which correspond to the E-G junction. The tip of the endoscope is placed at this level, which the surgeon marks with two clips. The intra-thoracic esophagus is mobilized by 9-12 centimeters to the level at which the left vagus nerve travels along the anterior aspect of the esophagus.

The distance between the E-G junction and the apex of the hiatus is measured after completely releasing the stomach, using an L-shaped instrument, which prevents errors associated with the two-dimensional video image. The upper arm of the L (90° based on the axis of the measurer) is placed at the apex of the diaphragm, and the distance between the base of the arm and the clip is measured in centimeters; the measurement is positive if the junction is above and negative if the junction is below the diaphragm. The length of the intra-abdominal portion of the esophagus that is suitable for the performance of a tension-free fundoplication is approximately 2.5 cm. If the E-G junction, with the stomach completely released, is still fixed above or astride the hiatus, the Collis technique is adopted. If the E-G junction is positioned below the hiatus by only 1-1.5 cm, a scenario in which even the application of slight downward traction on the stomach makes it possible to obtain the 2-3 cm of esophagus necessary to perform the fundoplication, its position creates a condition in which the decision of whether to perform a Collis gastroplasty becomes subjective. In such cases, the investigators generally perform the lengthening procedure if reflux symptoms have been present for many years, if the patient is obese, or if the patient is younger than 60 years. To perform the esophagus lengthening procedure, it is necessary to divide at least two short vessels. By turning the operating table toward the right side of the patient, the surgeon may simultaneously operate through the aforementioned 5 standard laparoscopic ports, as well as a left thoracoscopic port through which the instrument used to lengthen the esophagus is inserted. A thoracostomy is performed at the posterior axillary line at the V-VI-VII intercostal spaces, depending on the patient's body shape and size. A 12-mm valvular trocar may be used to prevent loss of pneumoperitoneum and to control intra-thoracic pressures.

The anesthesiologist passes a Maloney bougie 46 ch. into the esophagus and into the proximal stomach.

A no. 45 Endo GIA is inserted through the thoracic port; the tip of the instrument is delicately pressed against the left diaphragm to visually control the progression of the stapler from the port to the mediastinum. The stapler is fully visible through the hiatus as it penetrates the left mediastinal pleura. When it enters the abdominal cavity, the jaws are rotated toward the patient's left side.

The stapler is opened and positioned at the angle of His with its arms parallel but not too close to the Maloney bougie. To facilitate this maneuver and prevent the formation of a pouch between the suture lines and the angle of His, it may be necessary to pull the gastric fundus to the left when using the stapler.

The neo-esophagus is approximately 3 cm long. The mechanical suture line is covered with a sero- muscular running suture. A hiatoplasty is routinely performed; in the event of a type II-IV HH, the sutures applied to the diaphragmatic crura are reinforced with polytetrafluoroethylene-pledgeted sutures (two for each stitch, placed laterally at the edges of the crura and over the peritoneum). A floppy Nissen fundoplication (one 1.5-cm U stitch reinforced with pledgets) is performed. The superior edges of the fundoplication are placed above the clips, which mark the native E-G junction, to fully wrap the neo-esophagus. Two vertical U stitches intended to grab the inner, circular, muscular layer are applied laterally between the fundus and the esophagus to prevent slippage.

Follow-Up

Post-operatively, each of the patients participated in a free-of-charge outpatient follow-up program that entailed visits at 6 months, 12 months, and 2, 3, 4, and 5 years following surgery. At 1, 3, and 5 years, patients participated in a clinical interview and underwent both an upper GI endoscopy and a barium swallow study. The methodologies of these tests were the same as those used for the pre-operative work-up. Following the initial five-year follow-up period, patients were offered the opportunity to attend an outpatient clinical consultation every 3 years, as well as to undergo an endoscopy and a radiological examination of the esophagus and stomach. The follow-up procedures were established according to the "good practice criteria" accepted by the Italian Health Service. Patients voluntarily agreed to participate in the program. The length of the follow-up was calculated based on the amount of time that elapsed between the date of each patient's surgery and the day on which each patient appeared for the final follow-up visit.

An evaluation scale for the surgical results, from "excellent" to "poor" was used.

The results of cases in which a recurring HH was diagnosed by barium swallow, even an HH smaller than two centimeters, as well as those of cases in which medical therapy (H2 blockers or proton pump inhibitors) was necessary to control reflux symptoms or esophagitis, were classified as "poor".

ELIGIBILITY:
Inclusion Criteria:

Patients aged > 18 years with severe GERD symptoms and esophagitis associated with short esophagus

Exclusion Criteria:

Patients aged < 18 years Patients aged > 18 years with sliding hiatal hernia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 1995-01; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Number of patients with satisfactory results (Change from Baseline in the evaluation of symptoms and esophagitis at 12 months after surgery. | 12 months
  participants will be followed during the follow-up 12 months after surgery. 12 months after surgery the partecipants will perform clinical interview, upper gastrointestinal endoscopy and barium swallow

SECONDARY OUTCOMES:
Number of patients with satisfactory results | up to 60 months after surgery
  participants will be followed during the follow-up 60 months after surgery. 60 months after surgery partecipants will perform clinical interview, upper gastrointestinal endoscopy and barium swallow

CONTACTS AND LOCATIONS:
Overall Officials: Sandro Mattioli, MD, Principal Investigator — University of Bologna
Locations (1):
- Department of Medical and Surgical Sciences University of Bologna, Bologna, Bo, Italy

REFERENCES:
- [Derived] Lugaresi M, Mattioli B, Perrone O, Daddi N, Di Simone MP, Mattioli S. Results of left thoracoscopic Collis gastroplasty with laparoscopic Nissen fundoplication for the surgical treatment of true short oesophagus in gastro-oesophageal reflux disease and Type III-IV hiatal hernia. Eur J Cardiothorac Surg. 2016 Jan;49(1):e22-30. doi: 10.1093/ejcts/ezv381. Epub 2015 Oct 29. PMID 26518379
- See also: Department of Medical and Surgical Sciences University of Bologna — http://dimec.unibo.it